CLINICAL TRIAL: NCT04600778
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Cavosonstat Administered Twice Daily Compared With Placebo for 24 Weeks in Adult Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GSNOR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LVC-N91115-PS-II-01
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — cavosonstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): twice daily
  Interventions: Other: placebo
- Cavosonstat 5 mg (Experimental): twice daily
  Interventions: Drug: Cavosonstat 5 mg
- Cavosonstat 10 mg (Experimental): twice daily
  Interventions: Drug: Cavosonstat 10 mg
- Cavosonstat 25 mg (Experimental): twice daily
  Interventions: Drug: Cavosonstat 25 mg

INTERVENTIONS:
Other: placebo — placebo
  Arms: placebo
Drug: Cavosonstat 5 mg — Cavosonstat (low dose)
  Arms: Cavosonstat 5 mg
Drug: Cavosonstat 10 mg — Cavosonstat (medium dose)
  Arms: Cavosonstat 10 mg
Drug: Cavosonstat 25 mg — Cavosonstat (high dose)
  Arms: Cavosonstat 25 mg

SUMMARY:
Brief Summary: The purpose of this study is to to evaluate the efficacy and safety of Cavosonstat administered twice daily compared with Placebo for 24 Weeks in adult subjects with Chronic Obstructive Pulmonary Disease (COPD)

Detailed Description:To investigate the effect of cavosonstat compared with placebo, on the annualized rate of moderate-to-severe acute exacerbations of COPD (AECOPD) over 24 weeks of treatment.

To investigate:

1. The effect of cavosonstat compared with placebo, on the duration from baseline to first moderate AECOPD event
2. The effect of cavosonstat compared with placebo, on respiratory function, as assessed by post-bronchodilator percent-predicted forced expiratory volume in one second (ppFEV1)
3. The effect of cavosonstat compared with placebo on annualized rate of moderate AECOPD over 24 weeks of treatment
4. The effect of cavosonstat compared with placebo on annualized rate of severe AECOPD over 24 weeks of treatment
5. The safety and tolerability of cavosonstat compared with placebo
6. The pharmacokinetics of cavosonstat
7. Assessment of quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe COPD, who meet the following criteria (full details in main text):

  * Male or female aged between 40 and 75 years inclusive, at the time of informed consent
  * Patients with symptomatic COPD as defined by the 2019 GOLD diagnostic criteria
  * Post-bronchodilator (four puffs of albuterol) spirometry at screening demonstrating the following:

    1. FEV1/forced vital capacity (FVC) ratio of <0.70
    2. FEV1 ≥30% and FEV1 <80% of predicted normal
  * Current or prior history of ≥10 pack-years of cigarette smoking
  * Participants with COPD Assessment Test (CAT) score ≥10 at screening
  * Participants with a documented history of ≥1 moderate exacerbation within the year prior to screening
  * Participants with standard of care background therapy for three months and at a stable dose for at least one month, including either:
  * Single therapy: long-acting muscarinic agonist (LAMA), or
  * Double therapy: long-acting beta agonist (LABA) plus long-acting muscarinic agonist (LAMA) or inhaled corticosteroid (ICS) plus LABA or ICS plus LAMA, or
  * Triple therapy: LABA plus LAMA plus ICS
  * Meet the concomitant medication restrictions and continue to do so throughout the study
  * Have body mass index >21 kg/m2 and < 35 kg/m2
  * Males must agree not to donate sperm. They must be sexually abstinent or use a condom with all sexual partners. If the partner is of child-bearing potential, a condom with spermicide and a second reliable form of contraception must also be used
  * Females must be of non-childbearing potential, be sexually abstinent or use a highly effective form of contraception.
  * Able to sign an informed consent document

Exclusion Criteria:

* Patients meeting any of the following criteria must be excluded from the study (full details in main text):

  * Patients with other respiratory disorders: current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, uncontrolled or unstable sleep apnea, cor pulmonale, clinically significant pulmonary hypertension or other active pulmonary diseases
  * Chest X-ray (or computerized tomography [CT] scan) reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD
  * Moderate or severe AECOPD within the previous four weeks
  * An upper or lower respiratory tract infection that required the use of antibiotics within the previous four weeks
  * Long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for more than 12 hours a day
  * Oral therapies for COPD (e.g. oral steroids, theophylline and roflumilast) or antibiotics or oral corticosteroid therapy within four weeks prior to screening
  * Prior history of, or planned pneumonectomy or lung volume reduction surgery
  * Participation in the acute phase of a pulmonary rehabilitation program within four weeks of screening or planned during the study
  * History of malignancy of any organ system within five years, except skin cancer which has been stable over one year and the investigator believes is no clinical significance.
  * Patients with uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric, or ophthalmic diseases that the Investigator believes are clinically significant. This includes any hepatic disease or moderate to severe renal impairment.
  * Documented clinically significant cardiovascular disease such as: any history of arrhythmias, angina, recent (<1 year) or suspected myocardial infarction, congestive heart failure, unstable or uncontrolled hypertension, or diagnosis of hypertension within 3 months prior to Screening.
  * Known or suspected history of alcohol or drug abuse within the last 5 years. Positive urine drug screen and blood alcohol level screen.
  * Clinically significant abnormal values for laboratory safety tests (hematology, blood chemistry, viral serology or urinalysis) at Screening, as determined by the Investigator.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than twice the upper limit of normal.
  * Received an experimental drug within 30 days or five half-lives, whichever is longer.
  * Women who are pregnant or breast-feeding.
  * Prior exposure to a GSNOR inhibitor.
  * Major surgery (requiring general anesthesia) within 6 weeks prior to Screening, lack of full recovery from surgery at Screening, or planned surgery through the end of the study.
  * A disclosed history or one known to the Investigator, of significant non-compliance in previous investigational studies or with prescribed medications.
  * Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-02-03 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate-to-severe acute exacerbations of COPD | 24 weeks
  To investigate the effect of cavosonstat compared with placebo, on the annualized rate of moderate-to-severe acute exacerbations of COPD (AECOPD) over 24 weeks of treatment.